CLINICAL TRIAL: NCT07090447
Title: Evaluation of a Nutrition Education Guide for Patients With Chronic Liver Disease: Impact on the Patient and Caregiver
Brief Title: Evaluation of a Nutrition Education Guide for Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20.189
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cirrhosis
Keywords: nutrition education; cirrhosis; education strategy; nutrition guide
MeSH Terms: conditions — Fibrosis | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guide+ (Experimental): Participants who received and used the Nutrition in Cirrhosis guide
  Interventions: Behavioral: Nutrition in Cirrhosis guide
- Guide- (No Intervention): Participants who received standard of care

INTERVENTIONS:
Behavioral: Nutrition in Cirrhosis guide — Patients in the intervention group received a paper copy of the Nutrition in Cirrhosis guide and were instructed to read and use it over the 6 months study period. The Nutrition in Cirrhosis guide consists 7 chapters, namely:
  Chapter 1: Malnutrition - What is it and why is it so important?; Chapter 2: What should patients eat and what to avoid?; Chapter 3: Tips for when patients do not feel like eating; Chapter 4: Recipe list; Chapter 5: Using meal supplements; Chapter 6: Managing weight loss and cirrhosis; Chapter 7: What to expect in the hospital.
  Arms: Guide+

SUMMARY:
The goal of this prospective study is to evaluate the impact of the Nutrition in Cirrhosis guide in patients with chronic liver disease. Researchers compared the patients who received the Guide (Guide+ group) to the patients who received standard of care (Guide- group). Data collection occured at baseline, 3 and 6 months, and included evaluation of nutrition knowledge (questionnaire based on the Guide), quality of life (Chronic Liver Disease Questionnaire) and nutritional risk (Liver Disease Undernutrition Screening Tool). Satisfaction was evaluated with 3 focus groups including patients from the Guide+ group as well as a patient partner and thematic analysis was conducted.

DETAILED DESCRIPTION:
In this study, the investigators aimed to evaluate the impact of the Nutrition in Cirrhosis guide, an evidence-based educational resource created by a team of experts in Canada. The Guide was conceived in order to inform patients and help them follow nutritional guidelines for cirrhosis, which has been shown to be a challenge. Specifically, this study aimed to evaluate the impact of the Guide on patients' nutritional knowledge, quality of life and nutritional risk over a 6-month period, as well as changes in dietary intake. Secondly, the goal was to evaluate patients' satisfaction of the Guide using focus groups. In this randomized controlled mixed-methods study conducted at the Centre Hospitalier de l'Université de Montréal Research Center, patients in the intervention group (Guide+) received and used the Guide for 6 months, and a control group (Guide-) received standard of care. Data was collected at baseline, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* cirrhosis diagnosis documented by biopsy, radiological evidence, elastrography or decompensation event (such as hepatic encephalopathy, ascites and gastro-oesophageal bleeding)
* having access to Internet

Exclusion Criteria:

- non-french speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Nutritional knowledge | From enrollment to the end of intervention at 6 months
  The assessment of participants' nutritional knowledge was conducted using a questionnaire created by experts from the research team with the intent to be solely based on the chapters of the Guide. The questionnaire consists of 14 items related to nutritional recommendations (dietary intake, protein, sodium, etc.), as well as questions regarding nutritional choices in the context of cirrhosis, definitions of nutritional terms, food groups and nutrients.

SECONDARY OUTCOMES:
Health-related quality of life | From enrollment to the end of intervention at 6 months
  Patients' quality of life was assessed using the Chronic Liver Disease Questionnaire (CLDQ), a validated tool specific for patients living with chronic liver disease. This questionnaire consists of 29 items categorized into 6 domains: abdominal symptoms, activity, emotional function, fatigue, systemic symptoms, and worry. Each domain is scored on a scale from 1 (indicating severe impact) to 7 (indicating minimal impact), with higher scores reflecting a lower frequency of symptoms and, therefore, an improved health-related QoL. The overall score is obtained by calculating the average of the 29 items.
Nutritional risk | From enrollment to the end of intervention at 6 months
  The nutritional risk was evaluated using the Liver Disease Undernutrition Screening Tool (LDUST). The LDUST is an easy-to-use tool that allows patients to answer questions about the 6 components of the Malnutrition Identification Table, which is the consensus of the Academy of Nutrition and Dietetics and the American Society for Parenteral and Enteral Nutrition.
Dietary intakes | From enrollment to the end of intervention at 6 months
  Dietary intakes were assessed using a validated, web-based, self-administered 24h dietary recall (R24W) developed at Université Laval (Québec, Canada). Participants were invited by email to complete the R24W on 2 unannounced days (1 weekend day and 1 weekday) selected randomly by a computer algorithm over a 7-day period, at every data collection timepoint.
Satisfaction with the Guide | At the end of the 6-month intervention
  Three online focus groups were conducted between August 2022 and October 2024. To be eligible, participants had to be in the Guide+ group. Each focus group was of an average duration of one hour and included 2 to 4 patients along with a patient partner to ensure the patients felt at ease and to facilitate the discussion. Focus groups were conducted by the registered dietitian on the Zoom meetings platform. Discussions were semi-directed based on an interview Guide that was developed by the research team prior to sessions and approved by the ethics committee. The interview Guide covered various sections, namely patients' overall satisfaction, their opinion on the Guide's complexity and its daily applicability.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche du Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- See also: The Nutrition in Cirrhosis Guide — https://liver.ca/the-nutrition-in-cirrhosis-guide/